CLINICAL TRIAL: NCT03677648
Title: A Phase II Randomized, Placebo Controlled, Double-blind, Four Arms Dose-ranging Study to Evaluate the Efficacy and Safety of SHR0302 Compared to Placebo in Patients With Moderate to Severe Active Crohn's Disease
Brief Title: A Phase II Study in Patients With Moderate to Severe Active Crohn's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Reistone Biopharma Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RSJ10201
Record Dates: First submitted 2018-09-17; First posted 2018-09-19 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2022-06

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — ivarmacitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- SHR0302 dose A (Active Comparator): Participants randomized in this arm will receive dose A of SHR0302 until end of study at week 24.
  Interventions: Drug: SHR0302
- SHR0302 dose B (Experimental): Participants randomized in this arm will receive dose B of SHR0302 until end of study at week 24.
  Interventions: Drug: SHR0302
- SHR0302 dose C (Experimental): Participants randomized in this arm will receive dose C of SHR0302 until end of study at week 24.
  Interventions: Drug: SHR0302
- Placebo (Placebo Comparator): Participants randomized in this arm will receive placebo until week 12, and then will be re-randomized into one of the 3 active arms (dose A, dose B, and dose C of SHR0302) in a 1:1:1 allocation ratio until the end of study at week 24.
  Interventions: Drug: SHR0302; Drug: Placebos

INTERVENTIONS:
Drug: SHR0302 — The study drug, SHR0302, is designed to block the activity of an enzyme protein called JAK (known as a JAK inhibitor).
Drug: Placebos — Placebos
  Arms: Placebo

SUMMARY:
The proposed study is a randomized, double-blind, placebo-controlled, multi-center Phase II study to investigate the safety and efficacy of SHR0302 in patients with moderate to severe active Crohn's Disease. The study aims to evaluate the optimal dose of SHR0302 and time needed in inducing clinical remission in active CD. This is an 12+12 weeks study, in which participants who complete the first 12 weeks treatment phase, will have the option to enter a blinded active arms 12-week extension phase. Early withdrawn subjects during the first treatment phase cannot enter the extension phase. The total duration of the study participation, including extension and follow-up, will be approximately 26 weeks.

With the wealth of scientific evidence on JAK/STAT involvement in IBD, the data from similar class of new drugs and the current data on SHR0302 (JAK1 inhibitor), support the rationale to proceed with phase II studies to evaluate the efficacy and safety of SHR0302 in patients with moderate to severe active CD.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female subject at ≥18 and ≤ 75 years of age at randomization.
* Subjects with a documented three-month history of diagnosed ileal, colonic, or ileocolonic Crohn's Disease at the time of randomization.
* Currently having Crohn's Disease with Crohn's Disease Activity Index (CDAI) score ≥ 220 to ≤450.

Exclusion Criteria:

* Diagnosis of indeterminate colitis, or clinical findings suggestive of Ulcerative Colitis.
* Subject with CD with stoma, gastric or ileoanal pouch, proto-colectomy or total colectomy, symptomatic stenosis or stricture, history of bowel perforation, suspected abscess; actively draining fistula.
* Treatment naïve subjects diagnosed with Crohn's disease, (without previous exposure to treatment).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2019-05-14 (Actual); Primary Completion 2021-09-16 (Actual); Study Completion 2021-12-09 (Actual)

PRIMARY OUTCOMES:
The percentage of subjects achieving clinical remission at week 12. | week12
  The percentage of subjects achieving clinical remission at week 12, defined as Crohn's Disease Activity Index (CDAI) score < 150.

SECONDARY OUTCOMES:
The percentage of subjects achieving clinical remission defined as mean daily stool frequency (SF) ≤2.5, and abdominal pain (AP) ≤ 1 using the Patient Reported Outcome from CDAI at week 1, 4, 8, 12, 13, 16, and 24. | week 1, 4, 8, 12, 13, 16, and 24
  The percentage of subjects achieving clinical remission defined as mean daily stool frequency (SF) ≤2.5, and abdominal pain (AP) ≤ 1 using the Patient Reported Outcome from CDAI at week 1, 4, 8, 12, 13, 16, and 24.
The percentage of subjects achieving clinical remission defined as PRO2 < 8 at week 1, 4, 8, 12, 13, 16, and 24. | week 1, 4, 8, 12, 13, 16, and 24
  The percentage of subjects achieving clinical remission defined as PRO2 < 8 at week 1, 4, 8, 12, 13, 16, and 24.
The percentage of subjects achieving clinical response defined as a CDAI decrease from baseline of ≥ 100 points at week 1, 4, 8, 12, 13, 16, and 24. | week 1, 4, 8, 12, 13, 16, and 24
  The percentage of subjects achieving clinical response defined as a CDAI decrease from baseline of ≥ 100 points at week 1, 4, 8, 12, 13, 16, and 24.

CONTACTS AND LOCATIONS:
Overall Officials: Xiang Chen, Study Director — Reistone Biopharma
Locations (82):
- United States (6):
  - West Central Gastroenterology d/b/a Gastro Florida, Clearwater, Florida
  - Wellness Clinical Research, LLLC-Central Florida, Lake Wales, Florida
  - West Central Gastroenterology d/b/a Gastro Florida, Tampa, Florida
  - NECCR Primacare Research, LLC, Fall River, Massachusetts
  - Wilmington Health, Wilmington, North Carolina
  - Digestive Disease Specialists, Inc., Oklahoma City, Oklahoma
- China (36):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Yijishan Hospital of Wannan Medical College, Yingshan, Anhul
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Nanchang University, Guangzhou, Guangzhou
  - The Sixth Affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangzhou
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Tongji Hospital Affiliated to Tongji Medicine College, Huazhong University of Science & Technology, Wuhan, Hubei
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Henan Provincial People's Hospital, Pingxiang, Hunan
  - The First People's Hospital of Changzhou, Changzhou, Jiangsu
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - Wuxi People's Hospital, Wuxi, Jiangsu
  - Yangzhou First People's Hospital, Yangzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The first Hospital of Jilin University, Changchun, Jilin
  - Ruijin Hospital, Shanghai Jiaotong University, School of Medicne, Shanghai, Shanghai Municipality
  - Shanghai Xinhua Hospital, Shanghai, Shanghai Municipality
  - Shanghai East Hospital, Shanghai, Shanghai Municipality
  - Shanghai Changhai Hospital, Shanghai, Shanghai Municipality
  - Tianjin Union Medical Center, Tianjin, Tianjin Municipality
  - Sir Run Run Shaw Hospital, Affiliated with the Zhejiang University School of Medicine, Hangzhou, Zheijiang
  - Huzhou Central Hospital, Huzhou, Zheijiang
  - Nanfang Hospital of Southern Medical University, Changchun
  - Xiangya Hospital Central South University, Changsha
  - st China Hospital Sichuan University, Chengdu
  - Fujian Provincial Hospital, Fuzhou
  - Qilu Hospital of Shandong University, Jinan
  - Jiangsu Province Hospital, Nanjing
  - Nanjing First Hospital, Nanjing
  - The Affiliated Hospital of Nanjing University School, Nanjing
  - Renji Hospital, Shanghai Jiaotong University School of Medicine, Shanghai
  - The University of Hong Kong-Shenzhen Hospital, Shenzhen
  - Shanxi Provincial People's Hospital, Taiyuan
  - Second hospital of Shanxi Medical university, Taiyuan
- Poland (15):
  - Indywidualma Specjalistyczna Praktyka Lekarska Maciej Zymla, Knurów
  - Amicare Sp. z o.o. Sp.k, Lodz
  - SALVE Zakład Opieki Zdrowotnej Sp. zo.o., Lodz
  - Nzoz Allmedica Badania, Nowy Targ
  - Provita Profamilia, Piotrkow Trybunalski
  - SOLUMED Centrum Medyczne, Poznan
  - KO-MED Central Kliniczne Plulawy, Puławy
  - Gabinet Lekarski Bartosz Korczowski, Rzeszów
  - Specjalistyczna Praktyka Lekarska dr med. Marek Horynski, Sopot
  - KO-MED Centra Kliniczne Staszow, Staszów
  - EZ-MED Centrum Medyczne, Swidnica
  - Centrum Zdrowia MDM, Warsaw
  - Centralny Szpital Kliniczny MSW, Warsaw
  - Nzoz Vivamed, Warsaw
  - PlanetMed sp. z o.o., Wroclaw
- Ukraine (25):
  - RCI Chernivtsi Regional Clinical Hospital Dept of Gastroenterology Bukovinsky SMU, Chernivtsi
  - I.I.Mechnykov Dnipropetrovsk Regional Clinical Hospital, Dnipro
  - I.I.Mechnykov Dnipropetrovsk, Dnipro
  - Ivano-Frankivsk Hospital, Ivano-Frankivsk
  - Ivano-Frankivsk Med. University, Ivano-Frankivsk
  - CHI Kharkiv City Clinical Hospital #13, Kharkiv
  - Public nonprofit enterprise, Kharkiv
  - Kherson City Clinical Hospital, Kherson
  - Khmelnyski Regional Hospital, Khmelnytskyi
  - Tx-Dx Center Adonis Plus Ltd, Kiev
  - Healthy and Happy, Kyiv
  - Kyiv City Clinical Hospital, Kyiv
  - Kyiv Clin Hospital on Railway St. 2, Kyiv
  - Med. Cen.of Limited Liability, Kyiv
  - Kyiv Regional Hospital #2, Kyiv
  - Lviv Regional Clinical Hosp, Lviv
  - Communal City Clinical Hospital of Ambulance, Dept of Therapy #1 D.Halytskyi Lviv NMU, Lviv
  - Medical Center Pulse, Vinnytsia
  - RCH Vinnytsia, Dept. Therapy, Vinnytsia
  - Vinnytsia M I Pyrogov, Vinnytsia
  - CCH #1 Vinnytsia M.I. Pyrogov NMU Ch of Propaedeutics of IM, Vinnytsia
  - Communal Institution Center of the Primary Medical- Sanitary Care#2, Vinnytsia
  - Center of primary health care, Vinnytsia
  - City Clinical Hospital, Zaporizhzhya
  - O.F. Herbachevskiyi Zhytomyr Regional Clinical Hospital, Zhytomyr

IPD SHARING:
Plan to Share IPD: No